CLINICAL TRIAL: NCT01233778
Title: Canola and Flax Oils in Modulation of Vascular Function and Biomarkers of Cardiovascular Disease Risk
Brief Title: Canola Oil Multicentre Intervention Trial (COMIT)
Acronym: COMIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Collaborators: University of Manitoba (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: PKE COMIT
Record Dates: First submitted 2010-11-01; First posted 2010-11-03 (Estimated); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Cardiovascular Disease
Keywords: Cardiovascular disease; Omega-3 fatty acids; Inflammation; Endothelial function; Canola oil
MeSH Terms: conditions — Cardiovascular Diseases; Inflammation | interventions — Rapeseed Oil; Linseed Oil; Safflower Oil

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (5):
- Canola Oil (Experimental)
  Interventions: Dietary Supplement: Canola Oil
- High Oleic Acid Canola + DHA (Experimental)
  Interventions: Dietary Supplement: High Oleic Acid + DHA Canola Oil
- High Oleic Canola Oil (Experimental)
  Interventions: Dietary Supplement: High Oleic Acid Canola Oil
- Flax & Safflower Oil (60:40) (Experimental)
  Interventions: Dietary Supplement: Flax Oil
- Safflower & Corn Oil (75:25) (Experimental)
  Interventions: Dietary Supplement: Safflower Oil

INTERVENTIONS:
Dietary Supplement: Canola Oil — 60g Canola oil daily per 3000kcal diet provided in a supplemental shake
  Arms: Canola Oil
Dietary Supplement: High Oleic Acid + DHA Canola Oil — 60g high oleic acid canola oil + DHA daily per 3000kcal provided in a supplemental shake
  Arms: High Oleic Acid Canola + DHA
Dietary Supplement: High Oleic Acid Canola Oil — 60g high oleic acid canola oil daily per 3000kcal provided in a supplemental shake
  Arms: High Oleic Canola Oil
Dietary Supplement: Flax Oil — 36g flax oil + 24g safflower oil daily per 3000kcal provided in a supplemental shake
  Arms: Flax & Safflower Oil (60:40)
Dietary Supplement: Safflower Oil — 45g safflower oil + 15g corn oil daily per 3000kcal provided in a supplemental shake
  Arms: Safflower & Corn Oil (75:25)

SUMMARY:
The objectives of this study are to examine how the consumption of treatment oils (including canola oil, DHA enriched canola-oil, high oleic acid canola oil, flax oil, and safflower oil) influence endothelial function, inflammation, oxidation, body composition, and plasma lipoprotein characterization.

DETAILED DESCRIPTION:
The consequence of total fat consumption on circulating plasma lipids and the incidence of cardiovascular disease has long been a central theme in nutrition research. Less well known is the influence of specific fatty acids on vascular endothelial function and the oxidative and inflammatory responses characteristic of atherogenesis. Omega 3 ( ω-3) fatty acids, including plant derived alpha-linolenic acid (18:3n-3, ALA) and marine derived eicosapentaenoic (20:5n-3, EPA) and docosahexaenoic acid (22:6n-3, DHA) have been shown to effectively modulate multiple cardiovascular risk factors in epidemiological, animal model and human clinical investigations. ALA is most commonly consumed as a major component of dietary canola and flaxseed oils and has a recommended intake of 1.1 and 1.6 g/d for women and men, respectively. EPA and DHA are consumed as fatty fish or fish oil and algae supplements with current recommended intakes of 500 mg/d (combined EPA and DHA).

ALA is thought to improve cardiovascular health by modulating circulating lipid concentrations, altering membrane structure and function by enhancing the total ω-3 fatty acid content of cell membrane phospholipids, and reducing inflammatory reactions by blocking the formation of arachidonic acid derived eicosanoids. However, there are extensive knowledge gaps in our understanding of the molecular mechanisms and clinical efficacy of ω-3 fatty acids in human health and disease prevention. Therefore, the purpose of this study is to further examine these relationships.

Feeding protocol and study treatments:

The study will proceed as a double blind, randomized cross-over controlled feeding study. Each treatment phase will be 30 days in duration, separated by 4-week washout periods. Subjects will consume a fixed composition of a precisely controlled basal, weight-maintaining diet (35% energy from fat, 50% carbohydrate, and 15% protein) supplemented with 60g/d of the following treatment oils: 1) canola oil; 2) DHA enriched canola-oil; 3) high oleic acid canola oil; 4) flax/corn oil (40:60); or 5) safflower/corn oil (75:25). Study diets will be prepared in a metabolic kitchen facility at each clinical site. Three isocaloric meals will be prepared each day for every subject. A 7-day rotating menu cycle will be used. Subjects will consume at least 1 of 3 daily meals under supervision. The other meals will be prepared and packed for every subject to be taken out. The study control and intervention oils will be delivered in milkshakes provided twice daily. Subjects will be instructed to consume only the prepared meals and limit their intake of alcohol to 2 drinks/week and caffeinated calorie free beverages to 40oz (5 drinks) per day. Diets will be planned for every subject according to his/her energy requirements and will be nutritionally adequate.

ELIGIBILITY:
Inclusion Criteria:

* Aged 20-65 years
* BMI = 22-32 kg/m2

In addition, eligibility will be based on metabolic syndrome criteria where we define eligibility on the basis of subjects having elevated waist circumference + 1 or more of the remaining 5 criteria:

* Elevated waist circumference - > 102 cm for men and >88 cm for women
* Elevated triglycerides - ≥ 1.7 mmol/L ( ≥150mg/dl) ( no upper limit)
* Reduced HDL - < 1 mmol/L (<40 mg/dl) for men and < 1.3 mmol/L (<50 mg/dl)for women
* Fasting glucose - ≥ 100 mg/dl (no upper limit)
* Elevated blood pressure - systolic ≥130 and/or diastolic ≥85 mm HG

  * Unmedicated participants - upper limit of Stage 1 Hypertension: systolic ≤ 159 and/or diastolic ≤ 99 mm HG and participants must be free of end stage/target organ disease symptoms
  * BP medicated participants: acceptable as long as individuals meet the specified blood pressure range of <140/90 mmHg, and have been stable for at least 6 months.

Exclusion Criteria:

* Smokers**
* History of thyroid disease, diabetes, kidney or liver disease, heart disease, or other chronic diseases
* Heavy alcohol consumption (>14 drinks/week)
* Chronic anti-inflammatory medication use
* Lactation, pregnancy, or desire to become pregnant during the study
* Taking lipid lowering medications (cholestyramine, colestipol, niacin, clofibrate, gemfibrozil probucol, HMG CoA reductase inhibitors) within the last three months
* Not willing to refrain from blood/plasma donation during the study period
* Gall bladder removal

  * For purposes of the this study non-smoking is defined as >6 months smoke-free; there is some evidence to show that smoking cessation increases HDL levels and 6 months is adequate time for this to stabilize, however this time span was chosen based on the decreased rate of relapse after 6 months.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2010-10; Primary Completion 2012-03 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Endothelial Health | End of diet period 1 (week 4)
  Study subjects will undergo endothelial health assessment by EndoPAT analysis. The EndoPat procedure will occur while the subject is lying down in a relaxed state. Throughout the study, the inflation pressure of the EndoPAT device will be electronically set to 10mm Hg below diastolic BP. Testing begins with 10 min of rest. Following rest, baseline pulse amplitude is measured from each fingertip for 5 min. Next, arterial flow is interrupted for 5 min by a cuff placed on the forearm at an occlusion pressure of 250 mmHg. Following occlusion release, pulse amplitude recording continues for 5 min.
Endothelial Health | End of diet period 2 (week 12)
  Study subjects will undergo endothelial health assessment by EndoPAT analysis. The EndoPat procedure will occur while the subject is lying down in a relaxed state. Throughout the study, the inflation pressure of the EndoPAT device will be electronically set to 10mm Hg below diastolic BP. Testing begins with 10 min of rest. Following rest, baseline pulse amplitude is measured from each fingertip for 5 min. Next, arterial flow is interrupted for 5 min by a cuff placed on the forearm at an occlusion pressure of 250 mmHg. Following occlusion release, pulse amplitude recording continues for 5 min.
Endothelial Health | End of diet period 3 (week 20)
  Study subjects will undergo endothelial health assessment by EndoPAT analysis. The EndoPat procedure will occur while the subject is lying down in a relaxed state. Throughout the study, the inflation pressure of the EndoPAT device will be electronically set to 10mm Hg below diastolic BP. Testing begins with 10 min of rest. Following rest, baseline pulse amplitude is measured from each fingertip for 5 min. Next, arterial flow is interrupted for 5 min by a cuff placed on the forearm at an occlusion pressure of 250 mmHg. Following occlusion release, pulse amplitude recording continues for 5 min.
Endothelial Health | End of diet period 4 (week 28)
  Study subjects will undergo endothelial health assessment by EndoPAT analysis. The EndoPat procedure will occur while the subject is lying down in a relaxed state. Throughout the study, the inflation pressure of the EndoPAT device will be electronically set to 10mm Hg below diastolic BP. Testing begins with 10 min of rest. Following rest, baseline pulse amplitude is measured from each fingertip for 5 min. Next, arterial flow is interrupted for 5 min by a cuff placed on the forearm at an occlusion pressure of 250 mmHg. Following occlusion release, pulse amplitude recording continues for 5 min.
Endothelial Health | End of diet period 5 (week 36)
  Study subjects will undergo endothelial health assessment by EndoPAT analysis. The EndoPat procedure will occur while the subject is lying down in a relaxed state. Throughout the study, the inflation pressure of the EndoPAT device will be electronically set to 10mm Hg below diastolic BP. Testing begins with 10 min of rest. Following rest, baseline pulse amplitude is measured from each fingertip for 5 min. Next, arterial flow is interrupted for 5 min by a cuff placed on the forearm at an occlusion pressure of 250 mmHg. Following occlusion release, pulse amplitude recording continues for 5 min.

SECONDARY OUTCOMES:
Body Composition | Week 4, 12, 20, 28 and 36 - End of each diet period
  To assess regional changes in body fat deposition, subjects will undergo a dual energy X-ray absorptiometry (DXA) scan at baseline (beginning of study) and end of each intervention period. Waist circumference measurements also will be taken at this time to track how much fat is lost from the abdominal area of the body.
Production of long chain fatty acids | Week 4, 12, 20, 28 and 36 - End of each diet period
  On the 29th day of each diet phase you will be asked to consume three tablespoons of tagged water (known as deuterium). The movement of these tagged materials will allow us to assess the quantity of long chain fatty acids (EPA and DHA) that your body is producing in response to your diet. All of the above tagged materials are non-radioactive, non-toxic, and do not pose any health risk to you. Another fasting blood sample will be obtained when you return the next morning.
Plasma Lipids | Week 4, 12, 20, 28 and 36 - End of each diet period
  Twelve-hour fasting blood samples (30ml) will be collected on day 1, 2, 29 and 30 for analyses of plasma lipids. Blood samples obtained on day 1 and 2 will be used to measure baseline values for study endpoints, whereas blood samples obtained on the two last days will be used to measure final endpoint values.
Plasma Cytokines | Week 4, 12, 20, 28 and 36 - End of each diet period
  Twelve-hour fasting blood samples (30ml) will be collected on day 1, 2, 29 and 30 for analyses of C-reactive protein and inflammatory cytokines. Blood samples obtained on day 1 and 2 will be used to measure baseline values for study endpoints, whereas blood samples obtained on the two last days will be used to measure final endpoint values.

CONTACTS AND LOCATIONS:
Overall Officials: Penny M Kris-Etherton, PhD, RD, Principal Investigator — Penn State University
Locations (1):
- Penn State University, University Park, Pennsylvania, United States